CLINICAL TRIAL: NCT00101634
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-response Study to Evaluate the Efficacy and Safety of 3 Fixed Doses (25 mg eq, 50 mg eq, and 100 mg eq) of Paliperidone Palmitate in Patients With Schizophrenia
Brief Title: Efficacy and Safety of a Long Acting Anti-Psychotic Versus Placebo in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003562
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone palmitate; R092670; antipsychotic
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone palmitate

SUMMARY:
The purpose of this study is to determine the efficacy (how well the drug works), safety, and side effects of paliperidone palmitate compared to placebo in the treatment of the symptoms of schizophrenia in adults. The placebo used in this study was a nutritional substance known as 20% Intralipid emulsion given to patients requiring intravenous feedings.

DETAILED DESCRIPTION:
Many patients with schizophrenia have difficulty adhering to a daily oral treatment regimen. Long-acting injectable (LAI) formulations may provide therapeutic plasma concentrations over several weeks, thereby eliminating the need for daily oral medication and making compliance easier. This is a randomized (patients will be assigned to different treatment groups based solely on chance), double-blind (neither the patient nor the physician will know if placebo or drug is being given and at what dose), placebo-controlled, parallel group, multicenter, dose-response study in adults who have schizophrenia. The study consists of a screening period of no more than 7 days and a 13-week double-blind treatment period. The screening period includes 4 days for tolerability testing, if necessary. In the double-blind treatment period, patients will be randomly assigned to 1 of 4 treatment groups (3 fixed doses of paliperidone palmitate or placebo) to receive 4 i.m. injections of paliperidone palmitate or placebo on Days 1, 8, 36, and 64. The study, including the screening period, will last approximately 14 weeks. Efficacy will be assessed throughout the study using the Positive and Negative Symptom Scale for Schizophrenia (PANSS), the Clinical Global Impression-Severity (CGI-S), and the Personal and Social Performance Scale (PSP). Safety will be evaluated throughout the study by monitoring adverse events, extrapyramidal symptom (EPS) rating scales scores, clinical laboratory test results; vital signs and body weight measurements; electrocardiograms (ECGs); and physical examination findings. In addition, the tolerability of injections will be assessed. ER OROS paliperidone 3 mg/day for 4 days. Injections (i.m.) of paliperidone palmitate (25, 50, or 100 mg eq.) will be given on Days 1, 8, 36, and 64.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet diagnostic criteria for schizophrenia according to DSM-IV for at least 1 year
* meet PANSS score criteria
* have body mass index (BMI) of >15.0 kilogram(kg)/meter (m)2.

Exclusion Criteria:

* Patients who have primary active DSM-IV Axis I diagnosis other than schizophrenia
* have a decrease of >/=25% in the PANSS score
* have DSM-IV diagnosis of active substance dependence within 3 months of screening evaluation (nicotine and caffeine dependence are not exclusionary)
* have history of treatment resistance as defined by failure to respond to 2 adequate trials of different antipsychotic medications
* have any severe preexisting gastrointestinal narrowing (pathologic or iatrogenic)
* have significant risk of suicidal, homicidal or violent ideation or behavior
* current presence of any significant or unstable medication condition
* treatment with any protocol disallowed therapies
* clinically significant result from screening laboratory or ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2004-12; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change in total PANSS score from baseline to the end of the double blind treatment period.

SECONDARY OUTCOMES:
PSP and CGI-S scores from baseline to the end of of the double-blind treatment. Incidence of adverse events, labs and ECGs throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Efficacy and safety of 3 fixed doses of paliperidone palmitate versus placebo in patients with schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=530&filename=CR003562_CSR.pdf